CLINICAL TRIAL: NCT03073447
Title: Prospective Registry in Young Women Presenting Acute Myocardial Infarction in France: Clinical, Morphological and Biological Descriptive Analysis: WAMIF Study
Brief Title: WAMIF : Young Women Presenting Acute Myocardial Infarction in France
Acronym: WAMIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: French Federation of Cardiology (Other); I.V.S. Institut des Vaisseaux et du Sang (Unknown); Biosensors Europe SA (Industry); AstraZeneca (Industry); Boston Scientific Corporation (Industry); Abbott Medical Devices (Industry); Terumo Corporation (Industry); Daiichi Sankyo (Industry); Hexacath, France (Industry); Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-01
Record Dates: First submitted 2016-12-09; First posted 2017-03-08 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Acute Myocardial Infarction; Women Over 18 and Under 50 Years of Age
Keywords: Myocardial infarction; Women; Young; Primary PCI; Hormone
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- women under 50 years with acute MI (Other): this clinical study is to systematically pool clinical, morphological and biological data of young women (< 50 years) presenting an Acute MI and to assess their short-term (in-hospital) and mid-term (12 months) prognosis. The usual blood tests will be performed at the patient's admission and then repeated at least 24 hours after coronary angiography, including repeated sampling assays for troponin, in order to measure the peak, following the routine of the department The specific assays, corresponding to the tests carried out as part of the WAMIF study will be sampled before discharge.
  Interventions: Other: Specific blood sample of women under 50 years with acute MI

INTERVENTIONS:
Other: Specific blood sample of women under 50 years with acute MI — The specific assays, corresponding to the tests carried out as part of the WAMIF study will be sampled before discharge. Some assays, including hormonal and thrombophilia will be centralized in order to standardize the results and their interpretation. All the biological data will be pooled and analyzed by IVS. a sample of blood will be made for later analysis in the context of a serum bank.
  Other Names: specific assays

SUMMARY:
MI in elderly women seems to share the same pathophysiology than in men, especially plaque rupture associated with conventional risk factors. Therefore the questions is not solved on the pathophysiology and specific risk factors in young women whose prognosis is more severe. A complete descriptive analysis appears mandatory to understand the peculiarities, including not only morphological but also biological explorations as well.

To date no systematic descriptive analysis has been performed including clinical characteristics, cardiac and extra-cardiac morphological exploration and hormonal and immunological assays, particularly in young premenopausal women presenting MI.

This study will provide for the first time a complete analysis, including hormonal assays, never made in an "acute" population.

The main objective of this clinical study is to systematically pool clinical, morphological and biological data of young women (< 50 years) presenting an Acute MI and to assess their short-term (in-hospital) and mid-term (12 months) prognosis. The definition of MI is the one adopted in the Third definition published in 2012. As such an event occurs in a young patient, diagnostic and treatment may vary among centres. The incidence of such cases in each centre being low and practice inhomogeneous, no conclusion could be advanced concerning the study of associated, indeed predisposing factors.

The work aims to comprehensively and systematically collect all the clinical and laboratory data and the results of the all morphological explorations carried out during the care of these young women admitted for acute MI in high-volume centres.

No additional invasive act, without any direct benefit for the care of patients will be realized for research purposes.

All these examinations, in particular invasive morphological, are more and more integrated in the practice of modern interventional cardiology especially for complex or infrequent situations, like this setting. They afford accurate diagnosis of coronary disease on one hand and on the second hand they determine the causal or at least participating factor.

A comprehensive and systematic analysis of this particular entity that is MI in young woman, would improve our knowledge of this disease and then enable to offer patients a more appropriate treatment and monitoring. It is necessary to progress in the understanding of the mechanisms of the early onset of coronary artery disease in its most acute and most serious presentation and to clearly define the specificities of coronary disease in young women. Moreover, a more precise identification of risk factors of MI in a woman under 50 will allow a better screening and even introduction of preventive strategies.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death among women in France. In-hospital mortality after acute coronary syndrome (ACS) remains significantly higher than in men, with a relative risk of up to 150%, especially among young women1,2. Early mortality rate of myocardial infarction (MI) continues to decline but that of women remains higher.

Background The risk of ACS increases with age, especially after menopause and in the presence of classic cardiovascular risk factors such as hypertension or diabetes. Nevertheless premenopausal women presenting MI are not exceptional even in the absence of risk factors. The worse prognosis in women, particularly in individuals under 50 years could result from the combination of harsher clinical presentation, less typical symptoms, and delayed diagnosis. Moreover, it is not uncommon that an ACS occurs in young women without the usual risk factors. Hormonal changes in particular related to contraceptive treatments have been incriminated, likewise chronic inflammation related to systemic diseases. To date the impact of hormonal, inflammatory or thrombophilia changes has not been elucidated.

Nowadays use of endovascular imaging during diagnostic coronary angiography is become common practice in particular in the absence of obvious culprit thrombotic or obstructive lesion. These invasive imaging techniques such as intravascular ultrasound (IVUS) or OCT (Optical Coherence Tomography), bring highly relevant complementary information in this setting, particularly to clarify the mechanism of MI such as rupture or erosion of atherosclerotic plaque, spontaneous dissection or intramural hematoma. The incidence of these particular form of acute coronary artery lesions are higher in women, especially among the youngest one.

In young, an angioCT or angioMRI (aortic and/or cerebral) are often performed looking for other atherosclerotic risk locations or morphological abnormalities in favour of a particular disease such as a fibrodysplasia. PET scan (18FDGlusose scintigraphy), when available, provides a valuable complement: it is a functional imaging research for other arterial locations for hypermetabolic inflammatory arteritis.

Usual laboratory tests will be made at admission and discharge as done in routine practice. These tests include blood count, electrolytes, blood urea, creatinine, prothrombin time, activated partial thromboplastin time, glucose, HbA1C, lipide profil, hemoglobin electrophoresis, CRP, fibrinogen.

Moreover some tests are recommended in case of ACS in a young patient not made systematically. It is the objective of our work to make a comprehensive and systematic analyse. Some assays require special techniques, to avoid any variability and therefore bias in interpretation of results, those will be, after preparation of the samples in the original department, centralized: such as homocysteine, markers of thrombophilia and hormone assays. Individually, these markers have been associated with the presence and progression of atheroma. However, these assays are rarely made and have not been comprehensively and systematically studied in the population of young woman presenting MI.

Moreover it has long been accepted that women were less exposed than men to the risk of cardiovascular disease due to the protective role of oestrogen. However this assumption has been questioned by recent work on the hormonal treatment of menopause. The administration of oestrogen does not prevent ischemic arterial disease in postmenopausal women and may even be deleterious in older women. Then it then appears crucial to analyse hormone levels in the acute phase of MI in order to progress in the understanding of the hormonal role in ACS, so far this has never been made in this context.

Study design This is a prospective multicentric observational clinical study. All women under 50 years admitted in one of the 32 participating centres, for acute MI, with and without ST segment elevation, will be included.

Experimental plan

* For any women admitted for acute MI with or without ST segment elevation in an investigation centre, participation in the study will be proposed.
* Coronary angiography will be performed in emergency at admission according to current guidelines in case of STEMI. In case of NSTEMI, patients will benefit from coronary angiography according to defined risk stratification.
* An IVUS imaging will be done in centers that practice this technique, the data will be collected as part of the study. This imaging will be performed if possible during the initial coronary angiography in order to objectify intraluminal thrombus, plaque rupture, hematoma or spontaneous dissection. This diagnostic strategy is carried out in common practice in the participating centers in atypical situations, particularly in the absence of obstructive lesion or visible thrombus at angiography. OCT may be carried out in a second step after mechanical and/or pharmacological thrombectomy in order to improve sensitivity.
* Participation in the study will be proposed and agreement will be signed before discharge.
* In the centers performing cardiac MRI, the MRI data will be collected as part of the study. Cardiac MRI will be done at the earliest after coronary angiography during the same hospitalization.
* The usual blood tests will be performed at the patient's admission and then repeated at least 24 hours after coronary angiography, including repeated sampling assays for troponin, in order to measure the peak, following the routine of the department
* The specific assays, corresponding to the tests carried out as part of the WAMIF study will be sampled before discharge.
* During one of these blood samples a 5 ml sample of blood will be made for later analysis in the context of a serum bank.
* Some assays, including hormonal and thrombophilia will be centralized in order to standardize the results and their interpretation
* A second angiography associated with a challenge test by Methergin® can be planned, at the discretion of the referring cardiologist, within 5 days after the index event. This test will be especially recommended if no etiology has been found by OCT or MRI in order to diagnose a spastic angina. The test will be performed during coronary angiography with intravenous injection of 0.4 mg of Methergin® (méthylergotamine) followed by a control angiography 3 minutes followed by a test after intracoronary injection of nitrates.
* All the data will be collected locally with the help of clinical studies technicians from the WAMIF study
* All the biological data will be pooled and analyzed by IVS
* The data management will be performed by the clinical research assistant from the SFC
* A telephone interview will be conducted at 12 months to collect the major cardiovascular events (death from any cause, cardiovascular death, recurrent MI, stent thrombosis, stroke and major bleeding). These events will be specified through hospital reports.

Total study duration: 18 months + follow up at to 12 months: 30 months Inclusion period: 18 months Duration of participation for one patient: 12 months Number of participating centers: 32 Average number of inclusions per month per center: 0.5 to 1

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 and under 50 years of age
* Women admitted for MI defined by significant release of biological markers of myocardial necrosis associated with one of the following signs: chest pain and / or ECG abnormalities and / or loss of viable myocardium in imaging and / or thrombus to coronary angiography
* Coronary angiography performed
* Patient not objecting to the use of personal data.
* Beneficiary of a social protection (excluding AME)
* Signature of informed consentement form

Exclusion Criteria:

* Iatrogenic MI and those of patients who died before hospitalization
* Other causes of chest pain syndrome with elevated troponin, including myocarditis, Tako Tsubo, sepsis will be excluded after performing an MRI.
* Participation in other biomedical research protocol excluding registers
* Linguistic or mental disability or refusal to sign the informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
the combined endpoint of major cardiovascular events | From date of randomization until the date of first documented date of death from any cause, cardiovascular death, recurrent MI, stent thrombosis, stroke and major bleeding, whichever came first, assessed up to discharge of the patient
  The primary endpoint will be the combined endpoint of major cardiovascular events occurring during the index hospitalization: death from any cause, cardiovascular death, recurrent MI, stent thrombosis, stroke and major bleeding (defined as classified BARC 3 to 5).

SECONDARY OUTCOMES:
Anatomical characteristics of culprit lesions | from date of enrollment up to 12 months
  Anatomical characteristics of culprit lesions by intracoronary imaging techniques: part of erosions and plaque ruptures,
Frequency of the rare non atheromatous | through study completion, an average of 1 year
  Frequency of the rare non atheromatous forms such as spontaneous hematomas and dissections, coronary emboli, coronary spasms,
prevalence of classical cardiovascular risk factors | through study completion, an average of 1 year
  Precise prevalence of classical cardiovascular risk factors in this population
Presence or absence of a higher prevalence of diseases related to inflammation or thrombophilia | through study completion, an average of 1 year
  Presence or absence of a higher prevalence of diseases related to inflammation or thrombophilia
Influence of gynaecological and obstetrical status, hormonal parameters, and in particular hormonal profiles at risk: SHBG elevation | through study completion, an average of 1 year
  hormonal parameters, SHBG elevation will be measured
Number of extracardiac events | through study completion, an average of 1 year
  any extracardiac event will be reported
Prevalence of systemic diseases in this population, | through study completion, an average of 1 year
Prevalence of heredity | through study completion, an average of 1 year
Major cardiovascular events at 12 months after | through study completion, an average of 1 year
  Major cardiovascular events at 12 months after the index hospitalization: death from any cause, cardiovascular death, recurrent MI, stent thrombosis, stroke and major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane MANZO SILBERMAN, Principal Investigator — Hôpital LARIBOISIERE PARIS
Locations (29):
- France (29):
  - Chu Amiens Picardie, Amiens
  - Centre Hospitalier Annecy Genevois, Annecy
  - Centre Hospitalier D'Antibes Juan-Les-Pins, Antibes
  - Centre Hospitalier D'Argenteuil, Argenteuil
  - Centre Hospitalier D'Avignon, Avignon
  - CHU de Beauvais, Beauvais
  - Chru La Cavale Blanche, Brest
  - Hopital Louis Pasteur, Chartres
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu Dijon, Dijon
  - Chu Grenoble, Grenoble
  - Centre Hospitalier de Haguenau, Haguenau
  - Groupe Hospitalier de La Rochell, La Rochelle
  - Chru de Lille, Lille
  - Ch St Joseph St Luc, Lyon
  - Chu Hopital Nord, Marseille
  - Chu de Montpellier, Montpellier
  - Chu de Nimes, Nîmes
  - Centre Hospitalier Rene-Dubos, Paris
  - Hôpital LARIBOISIERE, Paris
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Hopital Europeen Georges-Pompidou, Paris
  - Hôpital Bichat-Claude Bernard, Paris
  - Chu de Rennes, Rennes
  - Chu de Rouen, Rouen
  - Clinique St Hilaire, Rouen
  - Hotel-Dieu Saint-Jacques, Toulouse
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Centre Hospitalier de Versailles, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manzo-Silberman S, Couturaud F, Bellemain-Appaix A, Vautrin E, Gompel A, Drouet L, Marliere S, Sollier CBD, Uhry S, Eltchaninoff H, Bergot T, Motreff P, Lahlou N, Cottin Y, Mounier-Vehier C, Gilard M, Montalescot G; WAMIF Investigators. Characteristics of Young Women Presenting With Acute Myocardial Infarction: The Prospective, Multicenter, Observational Young Women Presenting Acute Myocardial Infarction in France Study. J Am Heart Assoc. 2024 Oct;13(19):e034456. doi: 10.1161/JAHA.124.034456. Epub 2024 Sep 25. PMID 39319493